CLINICAL TRIAL: NCT02210910
Title: A Randomized, Two-arm, Prospective Study to Assess the Efficacy and Safety of InSpace™ Device Implanted Over a Rotator Cuff Repair in Comparison With Rotator Cuff Repair Only
Brief Title: InSpace™ System Over Rotator Cuff Repair in Comparison to Repair Alone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoSpace Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IS-CL-02-01
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Rotator Cuff Tear
Keywords: Massive Rotator Cuff Tear, Sub-acromial spacer, Best repair of rotator cuff
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Best Repair of torn Rotator Cuff (Sham Comparator): Subjects will undergo surgical intervention (usually arthroscopy) to perform debridement, acromioplasty if deemed necessary, long head of biceps tenotomy, and at least partial repair.
  Interventions: Procedure: Best Repair of torn Rotator Cuff
- InSpace™ system (Active Comparator): Subjects will undergo surgical intervention (usually arthroscopy) to perform debridement, acromioplasty if deemed necessary, long head of biceps tenotomy, and at least partial repair, and placement of the InSpace™ system.
  Interventions: Device: InSpace™ system over repair

INTERVENTIONS:
Device: InSpace™ system over repair
  Arms: InSpace™ system
Procedure: Best Repair of torn Rotator Cuff
  Arms: Best Repair of torn Rotator Cuff

SUMMARY:
This is a post-marketing study to further assess the safety and effectiveness of the InSpace™ in the study population in comparison to surgical RCT repair.

DETAILED DESCRIPTION:
The effectiveness will be assessed by comparing the scores of the ASES, Constant and Quick DASH outcome questionnaires with respect to pain reduction, improvement of activity of daily living (ADL) and improvement of range of motion (ROM).

ELIGIBILITY:
Main Inclusion Criteria:

* Age 40 or older.
* Positive diagnostic MRI of the affected shoulder indicating full thickness large to massive RCT of at least 3cm in diameter (according to Cofield classification2) involving one or more tendons. (MRI can be done up to 6 months prior to randomization.)
* Persistent pain and functional disability of the affected shoulder for at least 3 months.

Main Exclusion Criteria :

* Known allergy to the balloon material (copolymer of PLA and -θ-caprolactone).
* Evidence of significant osteoarthritis or cartilage damage in the shoulder
* Evidence of gleno-humeral instability
* Previous surgery of the shoulder in the past 2 years, excluding diagnostic arthroscopy
* Evidence of major joint trauma, infection, or necrosis in the shoulder
* Partial-thickness tears of the rotator cuff

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
The change in the Shoulder Score | baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel